CLINICAL TRIAL: NCT01015339
Title: A Randomized Multicenter Phase III Study Comparing Paclitaxel Plus Capecitabine With Capecitabine Maintenance Treatment or Cisplatin Plus Capecitabine in Metastatic Adenocarcinoma of the Stomach or Esophagogastric Junction
Brief Title: Paclitaxel Plus Capecitabine With Capecitabine Maintenance Treatment in Metastatic Adenocarcinoma of the Stomach or Esophagogastric Junction
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University (Other)
Collaborators: Roche Pharma AG (Industry)
Responsible Party: Principal Investigator, Shen Lin, M.D., Peking University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PAC-C; ML22697
Record Dates: First submitted 2009-11-17; First posted 2009-11-18 (Estimated); Last update posted 2015-05-19 (Estimated); Status verified 2015-05

CONDITIONS: Advanced Gastric Cancer
MeSH Terms: interventions — Paclitaxel; Capecitabine; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cisplatin plus capecitabine (Active Comparator)
  Interventions: Drug: capecitabine; Drug: cisplatin
- Paclitaxel plus Capecitabine (Experimental)
  Interventions: Drug: Paclitaxel; Drug: capecitabine

INTERVENTIONS:
Drug: Paclitaxel — 80mg/m2 infusion,d1,d8 every 3 weeks
  Arms: Paclitaxel plus Capecitabine
Drug: capecitabine — Dosing schedule: 1000mg/m2 bid, days 1-14, every 3 weeks
  Arms: Paclitaxel plus Capecitabine
Drug: capecitabine — Dosing schedule: 1000mg/m2 bid, days 1-14, every 3 weeks
  Arms: Cisplatin plus capecitabine
Drug: cisplatin — 80mg/m2, day 1 of every 3 weeks
  Arms: Cisplatin plus capecitabine

SUMMARY:
The purpose of this study is to investigate whether Paclitaxel Plus Capecitabine With Capecitabine Maintenance Treatment as 1st line treatment in he advanced gastric cancer is effective and safe.

ELIGIBILITY:
Inclusion Criteria:

* Having signed informed consent
* Age≥ 18 years old
* Histologically confirmed gastric adenocarcinoma
* Unresectable recurrent or metastatic disease
* Previous neo-adjuvant or adjuvant treatment for gastric cancer, if applicable, more than 6 months
* Previous chemotherapy with capecitabine or cisplatin, if applicable, more than 12 months.
* Measurable disease according to the RECIST criteria
* Karnofsky performance status ≥60
* Life expectancy of ≥2 month
* No prior radiotherapy except radiotherapy at non-target lesion of the study more than 4 weeks
* ALT and AST<2.5 times ULN (≤5 times ULN in patients with liver metastases)
* Serum albumin level ≥3.0g/dL
* Serum AKP < 2.5 times ULN
* Serum creatinine <ULN, and CCr < 60ml/min
* Bilirubin level < 1.5 ULN
* WBC>3,000/mm3, absolute neutrophil count ≥2000/mm3, platelet>100,000/mm3, Hb>9g/dl

Exclusion Criteria:

* Brain metastasis (known or suspected)
* Previous systemic therapy for metastatic gastric cancer
* Inability to take oral medication
* Previous therapy targeting at angiogenesis or vasculogenesis pathway or other targeted therapy
* Surgery (excluding diagnostic biopsy) within 4 weeks prior to study entry
* Contraindications of nuclear magnetic resonance image such as fitment of cardiac pacemaker , nerve stimulator, or aneurysm clip, and metallic foreign body in eye ball and so on.
* Allergic constitution or allergic history to protium biologic product or any investigating agents.
* Severe heart disease or such history as recorded congestive heart failure, uncontrolled cardiac arrhythmia, angina pectoris needing medication, cardiac valve disease, severe abnormal ECG findings, cardiac infarction , or retractable hypertension.
* Pregnancy or lactation period
* Any investigational agent within the past 28 days
* Other previous malignancy within 5 year, except non-melanoma skin cancer
* Previous adjuvant therapy with capecitabine+platinum,
* Pre-existing neuropathy>grade 1
* Legal incapacity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2009-11; Primary Completion 2015-08 (Estimated); Study Completion 2015-08 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | 3 year

SECONDARY OUTCOMES:
Tumor response rate | 1 year
Disease control rate | 1 year
Overall survival | 5 year
adverse evens | 5 year

CONTACTS AND LOCATIONS:
Overall Officials: Lin Shen, MD, Principal Investigator — Peking University, School of oncology, Department of GI oncology
Locations (1):
- Department of GI Oncology, Peking University, School of Oncology, Beijing, Beijing Municipality, China